CLINICAL TRIAL: NCT05461313
Title: Fully Constrained Acetabular Liner Versus Dual Mobility Hip Joint in the Surgical Treatment of Metastatic Bone Disease of the Hip - A Randomized, Open-Label, Two-Arm, Non-Inferiority Study Evaluating the Post-Operative Hip Dislocation Rate
Brief Title: Fully Constrained Acetabular Liner vs. Dual Mobility Hip Joint in the Surgical Treatment of Metastatic Bone Disease of the Hip
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Afrim Iljazi, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-21078128
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Cancer to the Hip
Keywords: Metastatic Bone Disease; Total Hip Arthroplasty; Hip Replacement; Constrained Liner; Dual Mobility; Orthopaedic Oncology
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Intervention Model Description: A Randomized, Open-Label, Two-Arm, Non-Inferiority Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constrained Liner (Other)
  Interventions: Other: Constrained Liner
- Dual Mobility Cup (Other)
  Interventions: Other: Dual Mobility

INTERVENTIONS:
Other: Constrained Liner — Subjects in this arm will receive a constrained liner with one of the following implants: Freedom Constrained Acetabular Liner (Zimmer Biomet), G7 Freedom Constrained Acetabular Liner (Zimmer Biomet) or Lubinus Acetabular Cup with a safety ring (LINK)
  Arms: Constrained Liner
Other: Dual Mobility — Subjects in this arm will receive a dual mobility cup with the following implant: Avantage Dual Mobility Cup (Zimmer Biomet)
  Arms: Dual Mobility Cup

SUMMARY:
The purpose of the current study is to investigate whether dual mobility liners are non-inferior til constrained liners regarding the post-operative hip joint dislocation risk following total hip replacement in patients with metastatic bone disease of the hip.

DETAILED DESCRIPTION:
The use of constrained liners in total hip arthroplasty (THA) in patients with metastatic bone disease of the hip (MBD) has increased at our department in recent years to avoid hip dislocation in this high-risk population. Hip surgeons seldom recommend the use of constrained liners in primary surgery due to the risk of polyethylene wear and high revision rates. An alternative to constrained liners are dual mobility cups, which have been shown to decrease the risk of dislocation in other high-risk THA operations such as revision THA and THA in hip fracture patients, while providing the added benefit of a less restricted range of motion of the joint. This study will investigate whether dual mobility cups are non-inferior to constrained liners regarding the post-operative joint dislocation risk in patients with MBD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with metastatic bone disease of the hip defined as bone lesions in the proximal femur because of secondary malignant growth of a primary cancer located elsewhere or bone lesions in the proximal femur due to hematological malignancies
* Determined eligible for total hip arthroplasty for metastatic bone disease of the hip and is planned to undergo surgery at the study site
* Provides informed consent prior to initiation of any study-specific activities/procedures

Exclusion Criteria:

* Previous osteosynthesis or endoprosthetic surgery of the ipsilateral hip
* Pelvic reconstruction of the ipsilateral hip
* Total femoral replacement of the ipsilateral femur
* It is not surgically viable to insert an acetabular cup and/or a femoral stem
* Subject is currently or has previously been enrolled in this study
* Subject is incapable of understanding the patient information or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative joint dislocation risk | 6 months
  The 6-months hip dislocation rate in patients receiving a dual mobility cup compared to patients receiving a constrained liner for the surgical treatment of MBD

SECONDARY OUTCOMES:
Post-operative joint dislocation risk | 3 months
  The 3-months hip dislocation rate in patients receiving a dual mobility cup compared to patients receiving a constrained liner.
Implant survival | 3 and 6 months
  The 3-months and 6-months implant survival in patients receiving a dual mobility cup compared to patients receiving a constrained liner.
Overall survival | 3 and 6 months
  The 3-months and 6-months overall survival in patients receiving a dual mobility cup compared to patients receiving a constrained liner.
Post-surgical and prosthesis related complications | 6 months
  The incidence of post-surgical and prosthesis-related complications in patients receiving a dual mobility cup compared to patients receiving a constrained liner. These include but are not limited to deep venous thrombosis, pulmonary embolism, wound infections, periprosthetic infections, periprosthetic fractures etc.
Karnofsky Performance Status Score | 3 and 6 months
  The 3-months and 6-months Karnofsky Performance Status Score in patients receiving a dual mobility cup compared to patients receiving a constrained liner and who are alive at the defined time point.
Musculoskeletal Tumor Society Score | 3 and 6 months
  The 3-months and 6-months MSTS in patients receiving a dual mobility cup compared to patients receiving a constrained liner and who are alive at the defined time point
Harris Hip Score | 3 and 6 months
  The 3-months and 6-months HHS in patients receiving a dual mobility cup compared to patients receiving a constrained liner and who are alive at the defined time point
European Quality of Life - 5 Dimensions Questionnaire | 3 and 6 months
  The 3-months and 6-months Eq-5d score in patients receiving a dual mobility cup compared to patients receiving a constrained liner and who are alive at the defined time point
Toronto Extremities Salvage Score for the lower extremity | 3 and 6 months
  The 3-months and 6-months TESS in patients receiving a dual mobility cup compared to patients receiving a constrained liner and who are alive at the defined time point

OTHER OUTCOMES:
Post-operative joint dislocation risk | 12 and 24 months
  The 1-year and 2-year hip dislocation rate in patients receiving a dual mobility cup compared to patients receiving a constrained liner.
Implant survival | 12 and 24 months
  The 1-year and 2-year implant survival in patients receiving a dual mobility cup compared to patients receiving a constrained liner.
Overall survival | 12 and 24 months
  The 1-year and 2-year overall survival in patients receiving a dual mobility cup compared to patients receiving a constrained liner.
Post-surgical and prosthesis related complications | 24 months
  The incidence of post-surgical and prosthesis-related complications in patients receiving a dual mobility cup compared to patients receiving a constrained liner. These include but are not limited to deep venous thrombosis, pulmonary embolism, wound infections, periprosthetic infections, periprosthetic fractures etc.
Karnofsky Performance Status Score | 12 and 24 months
  The 1-year and 2-year Karnofsky Performance Status Score in patients receiving a dual mobility cup compared to patients receiving a constrained liner and who are alive at the defined time point.
Musculoskeletal Tumor Society Score | 12 and 24 months
  The 1-year and 2-year MSTS in patients receiving a dual mobility cup compared to patients receiving a constrained liner and who are alive at the defined time point
Harris Hip Score | 12 and 24 months
  The 1-year and 2-year HHS in patients receiving a dual mobility cup compared to patients receiving a constrained liner and who are alive at the defined time point
European Quality of Life - 5 Dimensions Questionnaire | 12 and 24 months
  The 1-year and 2-year Eq-5d score in patients receiving a dual mobility cup compared to patients receiving a constrained liner and who are alive at the defined time point
Toronto Extremities Salvage Score for the lower extremity | 12 and 24 months
  The 1-year and 2-year TESS in patients receiving a dual mobility cup compared to patients receiving a constrained liner and who are alive at the defined time point

CONTACTS AND LOCATIONS:
Overall Officials: Afrim Iljazi, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Orthopedic Surgery, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Iljazi A, Sorensen MS, Weber KS, Villadsen A, Eriksson F, Petersen MM. Fully constrained acetabular liner vs. dual mobility hip joint in the surgical treatment of metastatic bone disease of the hip: study protocol for a randomized, open-label, two-arm, non-inferiority trial evaluating the post-operative hip dislocation rate. Trials. 2023 Mar 18;24(1):204. doi: 10.1186/s13063-023-07237-9. PMID 36934286